CLINICAL TRIAL: NCT07352449
Title: Investigation of the Acute Effects of Classical Abdominal Massage on Arterial Stiffness, Muscle Oxygenation, and Exercise Capacity in Patients With Chronic Constipation
Brief Title: Acute Effects of Abdominal Massage on Arterial Stiffness, Muscle Oxygenation and Exercise Capacity in Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gazi2709
Record Dates: First submitted 2025-12-08; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Constipation; Arterial Stiffness; Muscle Oxygenation
Keywords: chronic constipation; arterial stiffness; muscle oxygenation; exercise capacity
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: The study included 30 patients diagnosed with chronic constipation. Patients were randomly assigned to either the intervention group (n=15), which received a single 15-minute abdominal massage session, or the control group (n=15), which received no intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): All assessments in the study were completed in a single day before and after intervention. Arterial stiffness was assessed using the SphygmoCor XCEL device, exercise capacity using the 6-MWT, muscle oxygenation during the 6MWT using the Moxy® monitor, and quality of life using the Constipation Quality of Life Scale (CCQLS) and the modified Borg scale for defecation difficulty. Patients in the intervention group received a single 15-minute abdominal massage.
  Interventions: Other: Abdominal massage; Device: SphygmoCOR XCEL; Device: Moxy Monitor
- Control (Other): All assessments in the study were completed in a single day before and after intervention. Arterial stiffness was assessed using the SphygmoCor XCEL device, exercise capacity using the 6-MWT, muscle oxygenation during the 6MWT using the Moxy® monitor, and quality of life using the Constipation Quality of Life Scale (CCQLS) and the modified Borg scale for defecation difficulty. Patients in the control group received no intervention and were allowed to wait 15 minutes.
  Interventions: Device: SphygmoCOR XCEL; Device: Moxy Monitor

INTERVENTIONS:
Other: Abdominal massage — The intervention group received an abdominal massage performed by the researcher. During the massage, participants were placed in a supine position. The practitioner was positioned on the patient's left side, and all sessions were conducted by the same researcher to standardize the practice. A pillow was placed under the head, and the knees were slightly flexed if comfortable. The massage was performed clockwise, following the anatomical location of the intestines, on the abdominal wall. The duration of the massage was 15 minutes. The massage was initiated in the left lower quadrant of the sigmoid colon and continued throughout the entire abdominal region. Four basic manipulative movements were used in the intervention: superficial effleurage, deep effleurage, petrissage, and vibration. The treatment began with superficial petrissage (stroking) to relax the wall. Deep effleurage and petrissage maneuvers were then performed, and finally, the massage was concluded with vibration.
  Arms: Intervention
Device: SphygmoCOR XCEL — Arterial stiffness was assessed noninvasively with the SphygmoCor XCEL device, which has good validity and reliability in patients with chronic constipation . The device measured aortic systolic pressure (SBP), aortic pulse pressure (APP), augmentation pressure (AP), augmentation index (AIx), AIx normalized to 75 bpm (AIx@75), aortic diastolic pressure (DBP), aortic mean arterial pressure (MAP), aortic heart rate (HR) and ejection duration (ED).
Device: Moxy Monitor — Muscle oxygenation was measured using the "Moxy®" monitor (Moxy, Fortiori Design LLC, Minnesota, USA). The device was applied unilaterally to the dominant quadriceps femoris muscle during 6MWT.

SUMMARY:
Constipation is defined as having bowel movements fewer than three times per week or experiencing subjective complaints such as a sensation of incomplete evacuation, abdominal bloating, tightness, restlessness, or discomfort despite normal bowel frequency, while chronic constipation is not a disease but a symptom characterized by decreased defecation frequency, hard stools, straining, and a persistent feeling of incomplete evacuation, with its definition varying among individuals. The aim of the present study is to investigate the acute effects of a single session of classical abdominal massage on arterial stiffness, muscle oxygenation, exercise capacity, quality of life, and sleep quality in individuals with chronic constipation. At least 30 participants diagnosed with chronic constipation will be included and randomly allocated into an intervention group or a placebo group. In both groups, arterial stiffness, muscle oxygenation, exercise capacity, constipation-related quality of life, and sleep quality will be assessed. In the intervention group, all assessments will be conducted immediately before and after the massage session, whereas in the placebo group, assessments will be performed before and after a waiting period equivalent to the duration of the massage. Normality of the variables will be examined using the Shapiro-Wilk test, histograms, and detrended plots. For between-group comparisons at baseline, independent samples t-tests will be used for normally distributed variables and Mann-Whitney U tests for non-normally distributed variables, while categorical data will be compared using chi-square tests. Post-hoc comparisons will be conducted using Bonferroni-adjusted procedures, and the level of statistical significance will be set at p < 0.05.

DETAILED DESCRIPTION:
Constipation is a highly prevalent health problem that adversely affects physical, mental, and social well-being, thereby reducing health-related quality of life. In Türkiye, population-based studies indicate that its prevalence ranges widely across communities. Clinically, constipation is described as having fewer than three bowel movements per week or experiencing subjective symptoms such as incomplete evacuation, bloating, abdominal tightness, restlessness, and discomfort despite normal stool frequency. Its pathogenesis is multifactorial and influenced by dietary patterns, genetic predisposition, colonic motility and absorption, as well as behavioral, biological, and pharmacological factors. A sedentary lifestyle and inadequate fluid intake are recognized risk factors. Although various classification systems for constipation exist in the literature, the present study focuses specifically on individuals diagnosed with chronic constipation. Chronic constipation is not a disease in itself but a symptom characterized by reduced defecation frequency, hard stools, straining, and a persistent sense of incomplete evacuation, with its definition varying among individuals.

Physical activity is a lifelong behavior essential for maintaining and improving cardiorespiratory endurance, reducing obesity and related diseases, and promoting longevity. Multiple studies have shown a positive association between walking and bowel motility. Exercise, one of the structured components of physical activity, consists of planned, repetitive body movements aimed at improving one or more components of physical fitness, and has been reported to be negatively associated with chronic constipation in adults. In some populations, daily moderate-intensity exercise has been shown to substantially reduce constipation, although other findings suggest that its benefits may depend on symptom severity or age group. Reduced bowel motility is strongly linked to low levels of physical activity, and individuals with constipation often demonstrate decreased activity levels; consequently, a reduction in exercise capacity is also expected. However, no studies have directly examined exercise capacity in patients with chronic constipation. The current study aims to address this gap by investigating the effect of classical abdominal massage on exercise capacity in individuals with chronic constipation.

Constipation is also associated with cardiovascular events. Alterations in gut microbiota may contribute to atherosclerosis, elevated blood pressure, and cardiovascular complications. With increasing age, constipation frequently coexists with other cardiovascular risk factors. Straining during defecation can raise blood pressure and may precipitate events such as heart failure, arrhythmias, acute coronary syndromes, or even aortic dissection. Chronic constipation may also trigger psychological stress, potentially influencing blood pressure regulation. The Valsalva-like breathing pattern often observed during straining further supports this physiological relationship. Arterial stiffness, a marker of atherosclerosis, occurs due to thickening and loss of elasticity in arterial walls. The mesenteric arteries, which supply the small and large intestines, are anatomically positioned such that colonic displacement-common in constipated individuals-may impose tension on branches such as the superior mesenteric artery. Transverse colon ptosis can alter the anatomical orientation of the colon and its vascular supply, contributing to bowel dysfunction and worsening constipation. To date, no study has examined arterial stiffness in patients with chronic constipation, and the present research seeks to elucidate this relationship and explore the acute effects of classical abdominal massage on arterial stiffness.

Muscle oxygenation reflects oxygen delivery and utilization within target tissues as a consequence of metabolic respiration. As a key indicator of metabolic activity, muscle oxygen saturation (SmO₂) provides insight into muscular performance and the balance between oxygen supply and demand during rest and exercise. Efficient oxygen utilization is crucial for sustaining physical activity, yet no studies have investigated muscle oxygenation in individuals with chronic constipation. This study therefore also aims to determine the acute effects of classical abdominal massage on muscle oxygenation and to clarify the potential relationship between chronic constipation and altered tissue oxygen dynamics.

Quality of life is a multidimensional and highly individualized construct influenced by physical, psychological, social, economic, and cultural factors. Although constipation is not life-threatening, it imposes biological, psychological, sociocultural, and economic burdens that negatively affect an individual's quality of life. The bidirectional communication between the brain and the gastrointestinal system, mediated through neural and hormonal pathways, also involves feedback mechanisms that influence circadian rhythms and sleep regulation. Poor sleep can exacerbate gastrointestinal symptoms, while digestive disorders may disrupt sleep-wake cycles and reduce sleep quality. For this reason, the present study additionally explores the effects of classical abdominal massage on sleep quality and health-related quality of life.

A wide range of pharmacological and non-pharmacological treatments are used in the management of constipation. Due to the potential adverse effects and financial burden associated with laxatives, non-pharmacological approaches have gained notable importance. Abdominal massage is a safe, non-invasive method widely used in both healthy individuals and patients with constipation. Manual pressure applied to the abdominal wall may stimulate gas movement, enhance bowel sounds, increase peristaltic activity, and facilitate mechanical stimulation of digestive organs. Through techniques such as effleurage, petrissage, vibration, and tapotement, abdominal massage can reduce muscle tension, promote local circulation, enhance digestive function, stimulate gastric secretions, increase alertness and peristalsis, relieve constipation, and even reduce elevated blood pressure. The abdominal region's extensive fascial network allows massage to induce mechanical and reflex effects on the intestines by altering intra-abdominal pressure and applying force to the rectum. Physiological responses to massage encompass biomechanical, physiological, neurological, and psychological domains. Previous research has demonstrated the use of abdominal massage as a palliative technique for chronic constipation, fecal incontinence, abdominal muscle tone alterations, and abdominal pain, with no reported adverse effects. However, no prior study has investigated the acute effects of classical abdominal massage on arterial stiffness, muscle oxygenation, and exercise capacity in individuals with chronic constipation. The aim of the present study is to address this gap and provide novel insights into these physiological interactions.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18-65 years
* Clinically diagnosed with chronic constipation
* Willing and able to provide informed consent and voluntarily participate in the study

Exclusion Criteria

* Presence of cognitive impairment that may interfere with understanding questionnaire items or performing test instructions
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness (Aortic systolic pressure (SBP)) | First Day
  Aortic systolic pressure (SBP) was assessed noninvasively using the SphygmoCor XCEL system. This device estimates central (aortic) systolic blood pressure through a validated transfer function based on brachial cuff-derived waveforms. Measurements were performed in the supine position after an adequate rest period, in a quiet and temperature-controlled environment, according to the manufacturer's recommendations. The SphygmoCor XCEL has demonstrated good validity and reliability for the assessment of central hemodynamic parameters, including aortic SBP, in patients with chronic constipation.
Arterial stiffness (Aortic pulse pressure (APP)) | First Day
  Aortic pulse pressure (APP) was assessed noninvasively using the SphygmoCor XCEL system. APP was calculated as the difference between central aortic systolic pressure and central aortic diastolic pressure derived from brachial cuff-based waveform analysis using a validated transfer function. All measurements were performed with participants in the supine position after an adequate rest period, in a quiet and temperature-controlled environment, in accordance with the manufacturer's guidelines. The SphygmoCor XCEL has demonstrated good validity and reliability for the assessment of central hemodynamic parameters, including aortic pulse pressure, in patients with chronic constipation.
Arterial stiffness (Augmentation pressure (AP)) | First Day
  Augmentation pressure (AP) was assessed noninvasively using the SphygmoCor XCEL system. AP was defined as the absolute difference between the second and first systolic peaks of the central aortic pressure waveform, reflecting the contribution of wave reflection to central systolic pressure. Central aortic pressure waveforms were derived from brachial cuff-based measurements using a validated transfer function. All measurements were conducted with participants in the supine position following an adequate rest period, in a quiet and temperature-controlled environment, in accordance with the manufacturer's recommendations. The SphygmoCor XCEL has demonstrated good validity and reliability for the assessment of augmentation pressure in patients with chronic constipation.
Arterial stiffness (Augmentation index (AIx)) | First Day
  Augmentation index (AIx) was assessed noninvasively using the SphygmoCor XCEL system. AIx was calculated as the ratio of augmentation pressure to aortic pulse pressure and expressed as a percentage, reflecting the contribution of wave reflection to central arterial stiffness. Central aortic pressure waveforms were obtained from brachial cuff-based measurements using a validated transfer function. All measurements were performed with participants in the supine position after an adequate rest period, in a quiet and temperature-controlled environment, in accordance with the manufacturer's recommendations. The SphygmoCor XCEL has demonstrated good validity and reliability for the assessment of augmentation index in patients with chronic constipation.
Arterial stiffness (AIx normalized to 75 bpm (AIx@75)) | First Day
  AIx normalized to a heart rate of 75 beats per minute (AIx@75) was assessed noninvasively using the SphygmoCor XCEL system. AIx@75 was automatically calculated by the device using a validated algorithm that adjusts the augmentation index for heart rate, allowing standardized comparison between individuals. Central aortic pressure waveforms were derived from brachial cuff-based measurements using a validated transfer function. All measurements were performed with participants in the supine position following an adequate rest period, in a quiet and temperature-controlled environment, in accordance with the manufacturer's recommendations. The SphygmoCor XCEL has demonstrated good validity and reliability for the assessment of AIx@75 in patients with chronic constipation.
Arterial stiffness (Aortic diastolic pressure (DBP)) | First Day
  Aortic diastolic pressure (DBP) was assessed noninvasively using the SphygmoCor XCEL system. Central aortic diastolic pressure was derived from brachial cuff-based measurements using a validated transfer function applied to the recorded pressure waveforms. All measurements were performed with participants in the supine position after an adequate rest period, in a quiet and temperature-controlled environment, in accordance with the manufacturer's recommendations. The SphygmoCor XCEL has demonstrated good validity and reliability for the assessment of central aortic diastolic pressure in patients with chronic constipation.
Arterial stiffness (Aortic mean arterial pressure (MAP)) | First Day
  Aortic mean arterial pressure (MAP) was assessed noninvasively using the SphygmoCor XCEL system. Central aortic MAP was derived from brachial cuff-based measurements using a validated transfer function applied to the recorded pressure waveforms and calculated by the device according to standard hemodynamic principles. All measurements were performed with participants in the supine position after an adequate rest period, in a quiet and temperature-controlled environment, in accordance with the manufacturer's recommendations. The SphygmoCor XCEL has demonstrated good validity and reliability for the assessment of central aortic mean arterial pressure in patients with chronic constipation.
Arterial stiffness (Aortic heart rate (HR)) | First Day
  Aortic heart rate (HR) was assessed noninvasively using the SphygmoCor XCEL system. Heart rate was derived from the central aortic pressure waveform obtained through brachial cuff-based measurements using a validated transfer function. All measurements were performed with participants in the supine position after an adequate rest period, in a quiet and temperature-controlled environment, in accordance with the manufacturer's recommendations. The SphygmoCor XCEL has demonstrated good validity and reliability for the assessment of heart rate in patients with chronic constipation.
Arterial stiffness (Ejection duration (ED)) | First Day
  Ejection duration (ED) was assessed noninvasively using the SphygmoCor XCEL system. ED was derived from the central aortic pressure waveform and defined as the time interval between the onset of systolic upstroke and the end of systolic ejection, reflecting left ventricular ejection time. Central aortic pressure waveforms were obtained from brachial cuff-based measurements using a validated transfer function. All measurements were performed with participants in the supine position after an adequate rest period, in a quiet and temperature-controlled environment, in accordance with the manufacturer's recommendations. The SphygmoCor XCEL has demonstrated good validity and reliability for the assessment of ejection duration in patients with chronic constipation.
Muscle oxygenation | First Day
  Muscle oxygenation was measured using the "Moxy®" monitor (Moxy, Fortiori Design LLC, Minnesota, USA). The device was applied unilaterally to the dominant quadriceps femoris muscle during 6MWT.

SECONDARY OUTCOMES:
Exercise capacity | First day
  Functional exercise capacity was assessed with 6MWT according to the American Thoracic Society and European Respiratory Society criteria .
Assessment of Quality of Life | First Day
  Quality of life was assessed with the CCQLS. This self-report scale consists of 28 items and subscales of "worry/anxiety" (11 items), "physical discomfort" (4 items), "psychosocial discomfort" (8 items), and "satisfaction" (5 items). Each item is scored on a scale of 1 to 5. The total score ranges from 28 to 140, with higher scores indicating greater symptom severity or frequency, depending on the subscale, and worsening quality of life.
Heart rate (HR) | First day
  Heart rate (HR) was continuously monitored using a heart rate monitor during the 6-minute resting period, throughout the test, and during the recovery phase.
Blood pressure (BP) | First day
  Blood pressure (BP) was measured using a standard sphygmomanometer during the 6-minute resting period and in the recovery phase to assess hemodynamic responses.
Oxygen saturation (SpO₂) | First day
  Peripheral oxygen saturation (SpO₂) was continuously monitored using pulse oximetry during the 6-minute resting period, throughout the test, and during the recovery phase.
Respiratory rate (RR) | First day
  Respiratory rate (RR) was assessed manually by counting breaths per minute during the 6-minute resting period, throughout the test, and during the recovery phase.
Dyspnea | First day
  Perceived dyspnea was evaluated using the modified Borg scale (0-10), where 0 indicates no breathlessness and 10 indicates maximal breathlessness, during the 6-minute resting period, at the end of the test, and during the recovery phase.
Perceived exertion - body | First day
  Overall perceived exertion of the body was assessed using the modified Borg scale (0-10), where 0 represents no exertion and 10 represents maximal exertion, at the end of the test and during the recovery phase.
Perceived exertion - legs | First day
  Perceived exertion of the legs was evaluated using the modified Borg scale (0-10), where 0 represents no exertion and 10 represents maximal exertion, at the end of the test and during the recovery phase to assess localized muscular fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Yoleri, MSc, Study Chair — Gazi University; Meral Boşnak Güçlü, Prof, Study Director — Gazi University; Ramazan Kozan, MD, Principal Investigator — Gazi University; Musa Güneş, PhD, Principal Investigator — Karabük University; Elif Sıla Karaveli, Pt, Principal Investigator — Gazi University; Merve Bayrak, Pt, Principal Investigator — Gazi University; Zeyneb Süeda Kaledibi, Pt, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Cardiopulmonary Physiotherapy and Rehabilitation, Ankara, Çankaya 06490, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Birimoglu Okuyan C, Bilgili N. Effect of abdominal massage on constipation and quality of life in older adults: A randomized controlled trial. Complement Ther Med. 2019 Dec;47:102219. doi: 10.1016/j.ctim.2019.102219. Epub 2019 Oct 16. PMID 31780015
- [Result] Monteiro ER, Aguilera LM, Rua-Alonso M, Araujo GDS, Correa Neto VG, Bentes CM, Vilaca-Alves J, Reis VM, Ferreira AS, Marchetti PH, da Silva Novaes J. Effect of Manual Massage, Foam Rolling, and Strength Training on Hemodynamic and Autonomic Responses in Adults: A Scoping Review. Healthcare (Basel). 2025 Jun 7;13(12):1371. doi: 10.3390/healthcare13121371. PMID 40565397
- [Result] Supa'at I, Zakaria Z, Maskon O, Aminuddin A, Nordin NA. Effects of Swedish massage therapy on blood pressure, heart rate, and inflammatory markers in hypertensive women. Evid Based Complement Alternat Med. 2013;2013:171852. doi: 10.1155/2013/171852. Epub 2013 Aug 18. PMID 24023571
- [Result] Gibbons WJ, Fruchter N, Sloan S, Levy RD. Reference values for a multiple repetition 6-minute walk test in healthy adults older than 20 years. J Cardiopulm Rehabil. 2001 Mar-Apr;21(2):87-93. doi: 10.1097/00008483-200103000-00005. PMID 11314289
- [Result] Feldmann A, Schmitz R, Erlacher D. Near-infrared spectroscopy-derived muscle oxygen saturation on a 0% to 100% scale: reliability and validity of the Moxy Monitor. J Biomed Opt. 2019 Nov;24(11):1-11. doi: 10.1117/1.JBO.24.11.115001. PMID 31741352
- [Result] Nakagomi A, Shoji T, Okada S, Ohno Y, Kobayashi Y. Validity of the augmentation index and pulse pressure amplification as determined by the SphygmoCor XCEL device: a comparison with invasive measurements. Hypertens Res. 2018 Jan;41(1):27-32. doi: 10.1038/hr.2017.81. Epub 2017 Oct 5. PMID 28978987
- [Result] Honkura K, Tomata Y, Sugiyama K, Kaiho Y, Watanabe T, Zhang S, Sugawara Y, Tsuji I. Defecation frequency and cardiovascular disease mortality in Japan: The Ohsaki cohort study. Atherosclerosis. 2016 Mar;246:251-6. doi: 10.1016/j.atherosclerosis.2016.01.007. Epub 2016 Jan 13. PMID 26812003